CLINICAL TRIAL: NCT02226705
Title: Treatment of Rhino-Sinusal Mucormycosis Through Transnasal Endoscopic Surgery Extended to the Skull Base.
Brief Title: Endoscopic Surgical Treatment of Rhino-Sinusal Mucormycosis
Acronym: MICCA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: End of inclusion period
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P110151
Record Dates: First submitted 2014-07-25; First posted 2014-08-27 (Estimated); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Rhinocerebral Mucormycosis
Keywords: Rhinocerebral Mucormycosis; Surgery; Fungal Infection; Survival
MeSH Terms: conditions — Mycoses

STUDY DESIGN:
Intervention Model Description: Endoscopic surgical treatment
Oversight: Data Monitoring Committee: No

ARMS (1):
- Multiple Surgeries (Experimental): Patients undergoing transnasal endoscopic surgery
  Interventions: Procedure: Multiple transnasal endoscopic surgeries

INTERVENTIONS:
Procedure: Multiple transnasal endoscopic surgeries — Transnasal endoscopic surgery extended to the skull base

SUMMARY:
Radical endoscopic transnasal surgery associated with medical treatment with liposomal amphotericine B may increase the local control of Rhino-Sinusal Mucormycosis and the survival rate. The objective of this study is to evaluate the local control rate and survival rate at 3 months after radical endoscopic transnasal surgery extended towards the skull base in association with antifungal therapy and early surgical reevaluation of the extent of the disease.

DETAILED DESCRIPTION:
Introduction : Treatment of Rhino-Sinusal Mucormycosis remains a challenge because of the severity of the disease with high mortality rates. Mainly involving diabetic and immunodeficient patients, first clinical presentation is a common infection of the sinuses which can extend towards deep spaces of the face, orbits, the skull base and the brain. The mortality rates range from 20 to 50%, up to 80% in case of cerebral extension. through Transnasal Endoscopic Surgery extended to the Skull Base.

Hypothesis : We hypothesize that infected tissues are devascularized and because of that antifungal therapies can hardly reach areas of infected tissues. Radical endoscopic transnasal surgery associated with medical treatment with liposomal amphotericine B may increase the local control of the disease and the survival rate. Clinical evaluation of the extent of the disease within the first 7 days following initial surgery may represent a prognosis factor.

Methods :

First national mutlicentric and multidisciplinary cohort on Rhino-Sinusal Mucormycosis Radiological staging for evaluation of the extent of the disease using CT scan, MRI and PET Scan at initial stage before surgery Radical surgery and/or endoscopic transnasal surgery extended towards the skull base associated with liposomal amphotericine B medical treatment.

At day 7 new radiological evaluation and second surgical look to adapt surgical resection of infected tissues, perform biopsies to search for mycormycosis, biofilms and dosage of the concentration of liposomal amphotericin B inside tissues. New radiological and surgical looks in case of absence of local control obtained on the second look and further.

Study of the response rate by an endoscopic & scan follow-up (with biopsies for anatomopathological et mycological studies) at 1 month, 3 months, 6 months & one year. PET scan initially & at 3 months.

Number of subjects included : Phase II type trial (exclusion of a zero hypothesis of survival rate <50% ), N= 23 patients

Total length of the study 4 years Inclusion period time : 3 years Time of participation per patient : 1 year Number of center and/or participating departments: 24 Mean number of patients included per year and per center : 0 to 3 patients

ELIGIBILITY:
Inclusion Criteria:

* Man or woman, over 18 years old, presenting a mucormycosis on a sinus biopsy showing large filaments with non or little septae compatible with a mucoral or with a positive culture for a mucoral on a sinus sample associated to clinical head & neack anomalies (endoscopic) & scans compatible with a mucormycosis previous to the inclusion and this whatever the patient incumbent pathology.
* Patient treated by liposomal amphotericin B or just before being treated
* Signature of informed consent :

  * by the patient if he is able to express their will
  * by the family or close, if the patient is unable to consent
* Inclusion in emergency clause is possible ( CPP agreement ) if the patient is incapacitated , no close is present and that the surgery is urgent
* Person affiliated to a Health Security System (beneficiary)

Exclusion Criteria:

* Pregnancy, breastfeeding
* Disseminated Mucormycosis (involvment of one site distant from the head and neck)
* Known hypersensitivity to a polyene
* Absence of documentation of mucormycosis (histological, mycological)
* Contraindication to the completion of the surgery as provided in this protocol
* Patient is the subject of a guardianship or tutelage measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Local control rate and survival rate | 3 months
  To evaluate the local control rate and survival rate at 3 months after radical endoscopic transnasal surgery extended towards the skull base in association with antifungal therapy and early surgical reevaluation of the extent of the disease.

SECONDARY OUTCOMES:
Survival rates | 6 and 12 months
  Survival rates at 6 and 12 months
Study of the response rate | 1 and 3 months
  Study of the response rate at 1 and 3 months according to Segar criteria (Segal, Clin Infect Dis) using clinical, mycological and radiological evaluation.
Study of the local control | 3 months
  Study of the local control obtained at day 7+/-5 days and survival rate and response rate at 3 months.
Study of the association between local control and survival rate and response rate | 3 months
  Study of the association between local control obtained at 1 month and survival rate and response rate at 3 months.
Evaluation of the interest of CT PET scan | 3 months
  Evaluation of the interest of CT PET scan in studying clinical response at 3 months.
Radiological staging | 3 months
  Radiological staging: comparison of the initial extent of the mucormycosis at day 0 by CT scan and MRI and survival rate at 3 months and local control obtained at day 7.
Dosage of the amphotericin B concentration inside tissues | Day 7
  Dosage of the amphotericin B concentration inside tissues (infeusingcted and at the border of infected tissues) as obtained with biopsies at day 7.
Search for biofilms using confocal microscopy | Day 0 and Day 7
  Search for biofilms using confocal microscopy on infected tissues biopsies
Staging of sequellae | 3 months, 6 months and 1 year
  Staging of sequellae using quality of life questionnaires
Bank of mucormycosis tissues | Day 0, Day 7, Day 14, D21 and Day 28
  Bank of mucormycosis tissues at -80°C

CONTACTS AND LOCATIONS:
Overall Officials: Romain KANIA, PhD, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Lariboisière, Paris, France